CLINICAL TRIAL: NCT06601283
Title: Vitamin C Plus Cordyceps to Chemotherapy Related Anemia in Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-12
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Phytotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VC plus herbal medicine (Experimental): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks. Vitamin C 300 mg/day, TID, PO. Reishi, 2 g/day, BID, PO. Cordyceps, 2 g/day, BID, PO.
  Interventions: Drug: Vitmain C plus herbal medicine

INTERVENTIONS:
Drug: Vitmain C plus herbal medicine — nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks. Vitamin C 300 mg/day, TID, PO. Reishi, 2 g/day, BID, PO. Cordyceps, 2 g/day, BID, PO.

SUMMARY:
The purpose of this study is to evaluate the efficacy of low-dose vitamin C plus herbal medicine on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. The MPACT trial has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to gemcitabine combined with nab-paclitaxel including anemia, hand/foot numbness, fatigue, nausea, and malnutrition have impaired the tolerability of the regimen.

Vitamin C, also called ascorbate, is an essential nutrient for the human body. It modulates metabolism, immune reaction, collagen synthesis, and iron absorption. Some studies have shown that high-dose intravenous Vitamin C may be effective against various types of cancer. Meanwhile, medium or low dose of Vitamin C may enhance the tolerability of chemotherapy by increasing iron absorption, improving anemia, alleviating pain and hand/foot numbness, and thus improving quality of life for patients with pancreatic cancer. In addition, numerous evidence has proved the efficacy of Reishi and Cordyceps in alleviating the side effects related to chemotherapy.

The purpose of this study is to evaluate the efficacy of low-dose vitamin C plus herbal medicine (Reishi and Cordyceps) on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy. Fifty patients will be assigned to the experimental group (gemcitabine combined with nab-paclitaxel, Vitamin C, Reishi and Cordyceps). Rate of anemia, rate of hand/foot numbness, severity of pain, quality of life, and overall survival are measured.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to understand and the willingness to sign a written informed consent document.

  * Age ≥ 18 years and ≤ 80 years.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
  * Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
  * Adequate organ performance based on laboratory blood tests.
  * Presence of at least of one measurable lesion in agreement to RECIST criteria.
  * Hemoglobin (Hgb) ≥ 8 g/dL.
  * The expected survival ≥ 3 months.
  * Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* • Patients who have received anti-tumor treatment for other types of cancer in the last two years.

  * Patients who have received any form of anti-tumor therapy for pancreatic cancer.
  * The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
  * Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
  * Pregnant or nursing women.
  * Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
  * Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results, including active opportunistic infections or advanced (severe) infections, and diabetes that cannot be controlled after adequate clinical anti-hyperglycemia treatment according to guidelines, uncontrollable hypertension, cardiovascular disease (Class III or IV heart failure as defined by the New York Heart Association classification, congestive heart failure (CHF), myocardial infarction in the past 6 months , unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc).
  * Renal insufficiency or dialysis
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, nab-paclitaxel, or other agents used in the study.
  * Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
  * Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Rate of anemia | At the end of Cycle 1 (each cycle is 28 days)
  Rate of anemia after every cycle of chemotherapy

SECONDARY OUTCOMES:
Rate of Grade 3 neuropathy | At the end of Cycle 1 (each cycle is 28 days)
  Rate of Grade 3 neuropathy after every cycle of chemotherapy
Change of numeric rating scale, NRS | At the end of Cycle 1 (each cycle is 28 days)
  Change of NRS and the administration of analgesic drugs after every cycle of chemotherapy
Quality of life, QOL | At the end of Cycle 1 (each cycle is 28 days)
  Change of QOL after every cycle of chemotherapy
Overall survival，OS | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from randomization to the time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Das G, Shin HS, Leyva-Gomez G, Prado-Audelo MLD, Cortes H, Singh YD, Panda MK, Mishra AP, Nigam M, Saklani S, Chaturi PK, Martorell M, Cruz-Martins N, Sharma V, Garg N, Sharma R, Patra JK. Cordyceps spp.: A Review on Its Immune-Stimulatory and Other Biological Potentials. Front Pharmacol. 2021 Feb 8;11:602364. doi: 10.3389/fphar.2020.602364. eCollection 2020. PMID 33628175
- [Result] Sohretoglu D, Huang S. Ganoderma lucidum Polysaccharides as An Anti-cancer Agent. Anticancer Agents Med Chem. 2018;18(5):667-674. doi: 10.2174/1871520617666171113121246. PMID 29141563
- [Result] Wang X, Zhu X, Liu Y, Liu H, Xiao Z, Luo G. Efficacy of vitamin C on chemotherapy-related anemia in pancreatic cancer: study protocol for a randomized controlled trial. Trials. 2024 Jul 29;25(1):512. doi: 10.1186/s13063-024-08345-w. PMID 39075587